Official Title of the Study:

A Randomized Controlled Study Investigating the Effectiveness of Intravenous Dexamethasone Prophylaxis in Preventing Post-operative Urinary Retention in Spinal Anesthesia at Al-Makassed Hospital

**NCT Number: NCT07077850** 

Date of Document: 01/07/2025

## Al-Quds University Jerusalem Deanship of Scientific Research



جامعة القدس القدس سادة البحث العلمي

Research Ethics Committee Committee's Decision Letter

Date: June 14, 2025 Ref No: 385/REC/2025

Dears Dr. Mohammed Maree, Dr. Abeer Dar Hasan, Dr. Ahlam Hammoudeh, Dr. Islam Khairaldin, Dr. Majdi Abu Daoud, Dr. Mohammad Qino, Mr. Anas Barabrah, Mr. Tareq Jarrar, Ms. Sara Darawish, Ms. Baraah Farun,

Research ethics application. After reviewing your submission titled: "A Randomized Controlled Study Investigating the Effectiveness of Intravenous Dexamethasone Prophylaxis in Preventing Post-operative Urinary Retention in Spinal Anesthesia at Al-Makassed Hospital", the Research Ethics Committee (REC) at Al-Quds University confirms that your application aligns with our ethics guidelines, which are based on the principles outlined in the Declaration of Helsinki.

Please note that this approval does not replace other required permissions, such as for sample shipment or data sharing. We also request a copy of your final report or publication when available.

This approval is valid for one Year. If your research extends beyond this period, a renewal request will be necessary. The approval remains valid as long as there are no changes to the research protocol.

Sincerely,

Suheir Ereqat, PhD Associate Professor of Molecular Biology

Research Ethics Committee Chair

Cc. Prof. Hanna Abdel Nour - President Cc. Members of the committee

Cc. file

Abu-Dies, Jerusalem P.O.Box 20002

بوديس، القدس ص.ب. 20002 الفاد ، 201202 ، مركب

recearab@admin alanda ada